WALANT Versus Local Anesthesia in Central Venous Catheter Insertion

Unique Protocol Id: B.30.2.ATA.0.01.00/830

Document Date: 01.11.2023

INFORMED CONSENT FORM FOR ADULT PATIENTS

Research Project Title: Comparison of Wide-Awake Tourniquet-Free Local Anesthesia Technique (WALANT) and Local Anesthesia in Central Venous Catheter Insertion

Principal Investigator Name: Dr. Ayça ÇALBAY

Other Investigators Name: Assoc. Prof. Sultan Tuna AKGÖL GÜR, Assoc. Prof. Ümit ARSLAN, Research Assistant Dr. Muhammed Çağrı AYKUT, Research Assistant Dr. Murat Maksut ÇALBAY, Research Assistant Dr. Orhan Enes TUNÇEZ

You have been invited to participate in a study titled "Comparison of WALANT and Local Anesthesia in Central Venous Catheter Insertion." The reason for your invitation is that you need a chest tube. This study is being conducted for research purposes, and participation is voluntary. Before you decide to participate in the study, we would like to inform you about the research. After you have been fully informed about the study and your questions have been answered, you will be asked to sign this form if you wish to participate. This research is under the responsibility of Dr. Ayça ÇALBAY and Assoc. Prof. Dr. Ümit ARSLAN, both faculty members in the Department of Emergency Medicine and the Department of Thoracic Surgery at Atatürk University.

What is the purpose of the study? How many people, in addition to myself, will participate in this study?

The following information should be included under this heading:

- 1- The purpose of the study is to compare two different local anesthesia techniques that can be used in conscious, oriented/cooperative patients who require a central venous catheterization kit when presenting to the Emergency Department and Cardiovascular Surgery clinics.
- A total of 60 people are planned to participate in the study, including you.

What will I expect if I participate in this study?

The following information should be included under this heading:

- The methods used in the study will be used. The diagnostic, treatment, and intervention protocols that must be implemented from the moment you enter the emergency room or cardiovascular surgery clinic with complaints of shortness of breath will remain unchanged. The selection of available treatments will be based on your patient file number.
- Duration of the study

The study begins when your need for a chest tube is determined. It will end at the end of your treatment without affecting any steps in the required examination and treatment algorithm.

Are there any risks or discomforts associated with the study?

1. Pain may occur during the anesthetic treatment for central venous catheter insertion.

2. If you have an unknown allergy to the medications administered during local anesthesia or WALANT, you may experience an allergic reaction.

What are the benefits of participating in the study?

This study aims to identify a more comfortable local anesthesia method by minimizing pain for patients undergoing central venous catheterization.

How will my personal information be used? (This section will be kept as is)

Your study physician will use your personal information to conduct the study and statistical analyses, but your identity will be kept confidential. Ethics committees or official authorities may review your information only if necessary. You have the right to request information about your results at the end of the study. The study results may be published in the medical literature upon completion, but your identity will not be disclosed.